CLINICAL TRIAL: NCT06400030
Title: The Effects of BioCeramic Sealer With Single Cone Technique on the Healing of Periapical Lesions: A Randomized Controlled Trial
Brief Title: A Comparison Between Two Types of Sealers in the Healing of Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Endo-1-2024
Record Dates: First submitted 2024-04-20; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Periapical Lesions
Keywords: Single Cone Technique; Lateral Condensation; BioCeramic-based Sealer; AH Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AH Plus sealer Group (Control Group) (Other): in this group, root canal system was filled with AH Plus sealer in conjunction with lateral condensation.
  Interventions: Procedure: Root canal treatment with AH Plus sealer
- BioCeramic Sealer Group (Experimental Group (Experimental): in this group, root canal system was filled with BioCeramic-based sealer in conjunction with single gutta-percha cone.
  Interventions: Procedure: Root canal treatment with BioCeramic sealer

INTERVENTIONS:
Procedure: Root canal treatment with AH Plus sealer — - AH Plus sealer Group: the base and accelerator of AH Plus Sealer was mixed, then the walls of the canal were coated with the AH Plus sealer using K-File, then lateral condensation was performed through a number of gutta-percha cones.
  Arms: AH Plus sealer Group (Control Group)
Procedure: Root canal treatment with BioCeramic sealer — - BioCeramic Sealer Group: the canals in this group were filled using BioCeramic-based sealer and a single gutta-percha cone, and gently insert it into the root canal to the preselected working length without applying pressure.
  Arms: BioCeramic Sealer Group (Experimental Group

SUMMARY:
This clinical study will evaluate the effect of BioCeramic sealer with single cone compared with the control group treated with AH Plus with lateral condensation in root canal obturation on the healing of periapical lesions.

The study sample will consist of 41 patients with 65 teeth with clear periapical lesions.

Root canal obturation will be applied for all patients. BioCeramic sealer will be applied for the experimental group only.

The changes of the dimensions of the periapical lesion will be assessed using CBCT radiographs; pre- and post- treatment changes for each group will be evaluated individually.

DETAILED DESCRIPTION:
Periapical lesions is considered as the most common symptoms associated with infected root canals.

Recently, the BioCeramic sealer has been considered one of the most common endodontic sealer that possess antibacterial properties, so it can have an effective role in the healing of periapical lesions, as well as its ability to prevent periapical leakage due to its attachment to the dentinal walls and gutta-percha cones.

This study will evaluate the effect of BioCeramic sealer on the healing of periapical lesions and the changes of the dimensions of the lesions.

Root canal obturation with gutta-percha cones will be applied in the two groups: The control group will receive the AH Plus with lateral condensation technique, and the experimental group will receive BioCeramic sealer with single cone technique.

CBCT radiographs will be gotten before and after one year of the treatment to evaluate the periapical lesion dimensions changes.

ELIGIBILITY:
Inclusion Criteria:

* One maxillary anterior tooth with a clear periapical lesion at least.
* Normal anatomic features and straight or slightly curved roots.
* The treated teeth must have complete roots and a closed apex.
* The ability to isolate the teeth with a rubber dam and restore them.
* Good oral hygiene.
* Good systemic health.

Exclusion Criteria:

* Root caries.
* Root fractures or resorption.
* Signs of occlusal trauma on the treated tooth.
* Internal or external resorption.
* Active periodontal disease.
* Pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change in the periapical lesion diameter | before and after one year of the treatment (root canal obturation)
  This diameter of the periapical lesions is going to be measured on a CBCT image.
  Initially, the sections of the periapical lesions will be evaluated in the three planes (sagittal, coronal, and axial). The section that contains the largest area of the lesion in each studied plane, will be used for measurement.
  * If the shape of periapical lesion is circular, the periapical diameter would be taken (at this plane) relying on the scale in the program accompanying the radiograph (CBCT).
  * If the shape of periapical lesion is not circular, the largest and smallest diameter of the lesion will be taken (at this plane) depending on the scale in the program accompanying the CBCT image, then the mean diameter will be calculated by collecting the previous two diameter and dividing them by 2.
  Ultimately, the three diameters of the lesion (taken at the three planes) are collected and the total is divided into 3 to obtain the mean diameter of the lesion.

SECONDARY OUTCOMES:
Change in the presence of edema | before, after six months, and one year of the treatment (root canal obturation)
  The detection of the edema will be performed using clinical examination (palpating the buccal tissues of the treated tooth).
  Time Frame: before, after six months, and after one year of the treatment (root canal obturation)

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus University, Damascus, Syria

REFERENCES:
- [Background] Zavattini A, Knight A, Foschi F, Mannocci F. Outcome of Root Canal Treatments Using a New Calcium Silicate Root Canal Sealer: A Non-Randomized Clinical Trial. J Clin Med. 2020 Mar 13;9(3):782. doi: 10.3390/jcm9030782. PMID 32183124
- [Background] Martins JFB, Scheeren B, van der Waal SV. The Effect of Unintentional AH-Plus Sealer Extrusion on Resolution of Apical Periodontitis After Root Canal Treatment and Retreatment-A Retrospective Case-control Study. J Endod. 2023 Oct;49(10):1262-1268. doi: 10.1016/j.joen.2023.07.021. Epub 2023 Jul 28. PMID 37516239
- [Background] Chybowski EA, Glickman GN, Patel Y, Fleury A, Solomon E, He J. Clinical Outcome of Non-Surgical Root Canal Treatment Using a Single-cone Technique with Endosequence Bioceramic Sealer: A Retrospective Analysis. J Endod. 2018 Jun;44(6):941-945. doi: 10.1016/j.joen.2018.02.019. Epub 2018 Mar 29. PMID 29606401
- [Background] Khandelwal A, Janani K, Teja K, Jose J, Battineni G, Riccitiello F, Valletta A, Palanivelu A, Spagnuolo G. Periapical Healing following Root Canal Treatment Using Different Endodontic Sealers: A Systematic Review. Biomed Res Int. 2022 Jul 8;2022:3569281. doi: 10.1155/2022/3569281. eCollection 2022. PMID 35845966
- [Background] Del Fabbro M, Corbella S, Sequeira-Byron P, Tsesis I, Rosen E, Lolato A, Taschieri S. Endodontic procedures for retreatment of periapical lesions. Cochrane Database Syst Rev. 2016 Oct 19;10(10):CD005511. doi: 10.1002/14651858.CD005511.pub3. PMID 27759881